CLINICAL TRIAL: NCT00578877
Title: Contraceptive Effectiveness and Safety Study of the SILCS Diaphragm: the Pivotal Study
Brief Title: Contraceptive Effectiveness and Safety of the SILCS Diaphragm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); FHI 360 (Other); ReProtect Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CONRAD C05-103
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2017-08

CONDITIONS: Contraception
Keywords: Contraception; SILCS Diaphragm; Contraceptive Gel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Gynol II (2% N-9 gel)
  Interventions: Device: SILCS Diaphragm; Combination Product: Nonoxynol-9 Gel
- Arm 2 (Experimental): Buffer Gel
  Interventions: Device: SILCS Diaphragm; Combination Product: Buffer Gel

INTERVENTIONS:
Device: SILCS Diaphragm — SILCS Diaphragm used with 5 ml gel
Combination Product: Nonoxynol-9 Gel — Gynol II (2% N-9 gel)
  Arms: Arm 1
Combination Product: Buffer Gel — Buffer Gel
  Arms: Arm 2

SUMMARY:
This multi-center contraceptive effectiveness and safety study of the SILCS diaphragm will enroll approximately 450 couples at risk for pregnancy at six study sites in the U.S. The study will randomly assign approximately 300 couples to use the SILCS diaphragm with BufferGel and approximately 150 couples to use the SILCS diaphragm with Gynol II (2% N-9 gel). At two sites, a substudy involving colposcopy and microflora will be conducted in about 80 women (40 at each site). The primary objective of this study is to estimate the cumulative 6-month typical-use pregnancy probability for women using the SILCS diaphragm with a contraceptive gel.

DETAILED DESCRIPTION:
This multi-center contraceptive effectiveness and safety study of the SILCS diaphragm will enroll approximately 450 couples at risk for pregnancy w at six study sites in the U.S. The study will randomly assign approximately 300 couples to use the SILCS diaphragm with BufferGel (BG) and approximately 150 couples to use the SILCS diaphragm with Gynol II (2% N-9 gel). At two sites, a substudy involving colposcopy and microflora will be conducted in about 80 women (40 at each site). For certain evaluations, the data from a contraceptive study conducted by NICHD of the Ortho All-Flex diaphragm used with either BG or N-9 will be used as historical controls.

In the current study, each participant will agree to use the SILCS diaphragm with her assigned contraceptive gel as her only method of contraception for approximately 7 months (at least 190 days) and at least 6 menstrual cycles. Emergency contraception will be offered if unprotected intercourse occurs, according to local prescribing practices.

Each female participant will undergo four scheduled visits: Enrollment, After Cycle 1, After Cycle 3, and Final visits. Two weeks after enrollment, each participant will be called to determine if she has had any problems with the method and to assess compliance.

Recruitment for this study is expected to take about 12 months. Each subject's participation will last about 6-7 months. Site closeout is expected to take three months. The clinical portion of the study should last about 21 months. Data closure and analysis are expected to take three months and the Final Report two additional months.

ELIGIBILITY:
Female Inclusion Criteria

In order to enroll into the clinical trial, potential subjects must:

* be healthy sexually active women, at risk for pregnancy and desiring contraception;
* be within the age range of 18 through 40 years, inclusive;
* be at low-risk for HIV or STI infection, currently have (at least 4 months) a single sexual partner who is also at low-risk for HIV or STI infection, and expect the same partner for the study;
* have a negative urine pregnancy test ;
* have normal menstrual cycles with a usual length of 24 to 35 days over the last 2 months ;
* have a documented history of at least 6 weeks and two spontaneous, normal menstrual cycles since last pregnancy outcome, one spontaneous normal menstrual cycle after discontinuing hormonal contraception or therapy and 10 months since last DepoProvera injection;
* not be actively desiring pregnancy for approximately 7 months and willing to accept an unknown risk of pregnancy;
* be willing to engage in at least 4 acts of heterosexual vaginal intercourse per cycle ;
* be willing to be fitted with a standard diaphragm and use the SILCS diaphragm with assigned study gel during the study;
* be willing to only use the assigned study gel with the SILCS diaphragm as the sole method of contraception over the course of the study;
* agree not to participate in any other clinical trials during the course of the study;
* be willing and able to comply with study procedures and to return to the clinic for scheduled follow-up visits; and
* colposcopy and microflora substudy only:

  * be willing to avoid using tampons for 72 hours prior to clinic visits or any intravaginal product other than those provided by the investigator for the duration of participation; and
  * be willing to comply with substudy procedures. Male Criteria

The male partner must be at least 18 years old and must not:

* have a known fertility problem or vasectomy;
* have known risks for STIs including HIV:

  * have had more than one sexual partner in the past four months;
  * have shared injection drug needles within the past six months;
  * have had sex with a man within the past 12 months;
  * have, or suspected to have, HIV infection; or
  * have been diagnosed with or treated for any STI in the past six months;(with the exception of recurrent genital herpes or condylomata)
* have a known sensitivity or allergy to silicone, nylon, and/or spermicide or product containing N-9; and
* have taken an investigational drug or used an investigational device within 30 days prior to enrollment or previously participated in this study.

Female Exclusion Criteria

In order to enroll into the clinical trial, potential subjects must not:

* have an allergy to silicone, nylon, latex or dry natural rubber products, and/or spermicides or products containing N-9;
* have a history of toxic shock syndrome (TSS);
* have a suspected or diagnosed UTI or vaginitis, unless treated and symptoms resolved prior to enrollment;
* have a history suggestive of infertility, defined as any of the following:

  * known history of a fertility problem, sterilization, ectopic pregnancy, hospitalization for pelvic inflammatory disease (PID), or endometriosis unless participant has had a subsequent spontaneous intrauterine pregnancy; or
  * abnormalities on pelvic examination at enrollment that may impair fertility;
* have contraindications to pregnancy (medical condition) or chronic use of class D or X medications;
* have high risk for HIV or other sexually transmitted infections (STIs):

  * have had more than one sexual partner in the past four months;
  * have shared injection drug needles within the past six months;
  * have, or suspected to have, HIV infection; or
  * have been diagnosed or treated for any STI, including Trichomonas vaginalis, (with the exception of recurrent genital herpes or condylomata) or PID within the past six months prior to the enrollment visit;
* have signs or symptoms of current cervicitis, endometritis or PID or have clinical evidence of HSV on exam;
* be lactating or breastfeeding;
* have any abnormal vaginal bleeding or spotting within the month prior to enrollment;
* have any abnormal finding on pelvic examination which precludes her from participating in the trial;
* have had a vaginal or cervical biopsy within one week or vaginal surgery within the three months prior to enrollment;
* have an abnormal Pap smear in the past 12 months defined as:

  * ASC-US without a normal repeat Pap smear at least 6 months later;
  * ASC-US with positive reflex high-risk HPV testing (ASC-US/HPV+) or LSIL except when a colposcopy was performed (with or without biopsy) and found no evidence of high-grade disease (CIN II or worse) unless treatment is indicated per local standard of care;
  * ASC-H, atypical glandular cells, or HSIL unless treatment was received and follow-up at least 6 months after the treatment showed no evidence of disease;
  * malignant cells;
* consume (on average) greater than 3 alcoholic beverages per day;
* have a past (within 12 months) or current history of drug abuse ;
* have previously participated in or completed this study;
* have a vaginal or cervical anatomic abnormality that would interfere with the proper placement and retention of the device;
* have other conditions that would constitute contraindications to participation or would compromise ability to comply with the study protocol;
* have taken an investigational drug or used an investigational device within the past 30 days; and
* have deep epithelial disruption on colposcopic exam (SUBSTUDY).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Frezieres, MSPH, Principal Investigator — Californial Family Health Council, Inc; Mitch M Creinin, MD, Principal Investigator — University of Pittsburgh; Lynn Bradley, M.Sc., Principal Investigator — John Hopkins Community Physicians; David Archer, MD, Principal Investigator — Eastern Virginia Medical School; Alfred Poindexter, MD, Principal Investigator — Advances in Health, Inc.; Kurt Barnhart, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - California Family Health Council, Inc, Los Angeles, California
  - John Hopkins Community Physicians, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Advances in Health, Inc., Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Derived] Schwartz JL, Weiner DH, Lai JJ, Frezieres RG, Creinin MD, Archer DF, Bradley L, Barnhart KT, Poindexter A, Kilbourne-Brook M, Callahan MM, Mauck CK. Contraceptive efficacy, safety, fit, and acceptability of a single-size diaphragm developed with end-user input. Obstet Gynecol. 2015 Apr;125(4):895-903. doi: 10.1097/AOG.0000000000000721. PMID 25751199

RESULTS

PARTICIPANT FLOW:
Groups:
- N-9 Gel With SILCS Diaphragm: Participants used the SILCS diaphragm with the N-9 gel as her only method of contraception for at least 190 days and at least 6 menstrual cycles
- BufferGel With SILCS Diaphragm: Participants used the SILCS diaphragm with BufferGel as her only method of contraception for at least 190 days and at least 6 menstrual cycles
Period: Overall Study
Arm/Group | N-9 Gel With SILCS Diaphragm | BufferGel With SILCS Diaphragm
Started | 150 | 300
Completed | 69 | 172
Not Completed | 81 | 128
Not completed — Lost to Follow-up | 8 | 10
Not completed — early discontinue | 61 | 101
Not completed — did not provide follow-up data | 12 | 17

BASELINE CHARACTERISTICS:
Population: treated population who answered the item
Groups:
- Total: Total of all reporting groups
Arm/Group | N-9 Gel With SILCS Diaphragm | BufferGel With SILCS Diaphragm | Total
Number analyzed (Participants) | 138 | 283 | 421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 283 | 421
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6) | 28.7 (6.0) | 28.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 283 | 421
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 138 | 283 | 421

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Pregnancy Among Users of the SILCS Diaphragm Used With Contraceptive Gel Over 6 Months of Typical Use
Time Frame: 6 months
Measure: Number; unit: percent probability
Arm/Group | N-9 Gel With SILCS Diaphragm | BufferGel With SILCS Diaphragm
Number analyzed (Participants) | 138 | 283
percent probability | 12.5 | 9.6

2. Secondary Outcome: Percent Women With Urogenital Adverse Events.
Description: Clinically evaluate the safety of the SILCS diaphragm used with contraceptive gel over 6 months of use.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | N-9 Gel With SILCS Diaphragm | BufferGel With SILCS Diaphragm
Serious Adverse Events (participants affected / at risk) | 1/137 | 3/278
Other Adverse Events (participants affected / at risk) | 85/137 | 179/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-9 Gel With SILCS Diaphragm (N=137) | BufferGel With SILCS Diaphragm (N=278)
Intentional Suicide (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post Surgical Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-9 Gel With SILCS Diaphragm (N=137) | BufferGel With SILCS Diaphragm (N=278)
Abnormal vaginal bleeding (Reproductive system and breast disorders) | 21 (21) | 38 (38)
Pain, irritation, pruritus (Reproductive system and breast disorders) | 48 (48) | 104 (104)
Symptomatic vaginal infection (Reproductive system and breast disorders) | 16 (16) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data obtained from a clinical trial in which 2 or more research centers participate cannot be published or presented by any of the individual investigators before the end of the clinical trial. Only after publication of the pooled results can data from individual centers be published.

When the Principal Investigator wishes to write a paper using data collected from his or her own center, the Recipient Institution agrees to allow CONRAD and USAID the opportunity to review & provide comments.